CLINICAL TRIAL: NCT02696265
Title: Complex Fractionated Atrial Electrocardiograms (CFAEs) Spatiotemporal Dispersion Guided Ablation Versus Pulmonary Vein Isolation (PVI) Guided Ablation in Persistent Atrial Fibrillation, a Multicenter Randomized Trial
Brief Title: CFAE/Spatiotemporal Dispersion Guided Ablation Versus PVI Guided Ablation in Persistent AF
Acronym: CIPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diagram B.V. (Other)
Collaborators: Biosense Webster, Inc. (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9227; 15.09159 (Other: Ethical Committee)
Record Dates: First submitted 2016-02-18; First posted 2016-03-02 (Estimated); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Chronic Atrial Fibrillation
Keywords: Atrial Fibrillation; Complex Fractionated Atrial Electrocardiograms; Pulmonary Vein Isolation; Ablation; CFAE/spatiotemporal dispersion guided ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CFAE guided ablation (Active Comparator): CFAE/spatiotemporal dispersion guided ablation: CFAE mapping and ablation during AF aimed at restoring sinus rhythm during ablation.
  Interventions: Procedure: CFAE guided ablation
- PVI guided ablation (Active Comparator): PVI guided ablation: wide antral pulmonary vein isolation during mapping catheter control of pulmonary vein signals.
  Interventions: Procedure: PVI guided ablation

INTERVENTIONS:
Procedure: CFAE guided ablation — CFAE/spatiotemporal dispersions mapping and ablation during AF aimed at restoring sinus rhythm during ablation. Pulmonal vein isolation will be checked before and after ablation using a mapping catheter.
  Arms: CFAE guided ablation
Procedure: PVI guided ablation — Wide antral pulmonary vein isolation during mapping catheter control of pulmonary vein signals
  Arms: PVI guided ablation

SUMMARY:
Objective: The purpose of this study is to compare the efficacy and safety of ablation of Atrial Fibrillation (AF) drivers marked by spatiotemporal dispersions and Complex Fractionated Atrial Electrocardiograms (CFAEs) to Pulmonary Vein Isolation (PVI) based ablation in patients with persistent AF.

Hypothesis: CFAE/spatiotemporal dispersion guided ablation will increase AF free survival compared to a PVI guided ablation.

Patient population: Patients with persistent AF will be randomized based on a 2:1 ratio into one of two study arms:

* CFAE/spatiotemporal dispersion guided ablation: CFAE mapping and ablation during AF aimed at restoring sinus rhythm during ablation.
* PVI guided ablation: wide antral pulmonary vein isolation during mapping catheter control of pulmonary vein signals

DETAILED DESCRIPTION:
Design: A prospective, multicenter, randomized unblinded clinical study.

Objective: The purpose of this study is to compare the efficacy and safety of ablation of AF drivers marked by spatiotemporal dispersions and CFAEs guided ablation to PVI guided ablation in patients with persistent AF.

Hypothesis: CFAE/spatiotemporal dispersion guided ablation will increase AF free survival compared to a PVI guided ablation.

Enrollment: 180 patients will be enrolled in this study.

Clinical Sites: International (including non EU-countries), multicenter study.

Patient population: Patients with persistent AF (defined as atrial fibrillation which is sustained beyond 7 days but no more than one year, or lasting less than 7 days but necessitating pharmacologic or electrical cardioversion, but lasting longer than 48 hours) should be documented either on 12-lead ECG, transtelephonic monitoring (TTM), ambulatory holter monitoring (HM) or telemetry strip and a physician's note showing continuous AF. Furthermore patients who have failed at least one Anti Arrhythmic Drug (AAD) (Class I or III) as evidenced by recurrent symptomatic AF or intolerable side effects of the AAD. Eligible patients who sign the study informed consent form will be randomized based on a 2:1 ratio into one of two study arms:

* CFAE/spatiotemporal guided ablation: CFAE/spatiotemporal dispersion mapping and ablation during AF aimed at restoring sinus rhythm during ablation. Pulmonal vein isolation will be checked before and after ablation using a mapping catheter
* PVI guided ablation: wide antral pulmonary vein isolation during mapping catheter control of pulmonary vein signals

Primary Endpoint: Freedom from recorded AF or atrial flutter or atrial tachycardia recurrences (>30 seconds) without the use of AADs through 18 months follow-up, post-blanking, on either a 12 lead ECG on visits or on 24 hour holter monitoring or on symptom driven event monitoring.

CFAE/spatiotemporal dispersions procedural details: To increase the accuracy of CFAE mapping, the Pentaray mapping catheter will be used to define spatiotemporal dispersion areas of CFAEs as specific targets of ablation as described by Seitz (see also citation) as follows. Dispersion areas are defined as clusters of electrograms, either fractionated or non-fractionated, that display interelectrode time and space dispersion at a minimum of 3 adjacent bipoles such that activation spread over all the AFCL. At each bipole in a dispersion area, one or more of the following fractionated or nonfractionated electrogram morphologies can be found:

1. continuous, low-voltage fractionated electrograms ("continuously fractionated signal");
2. bursts of fractionated electrograms ("trains of fractionation");
3. fast nonfractionated electrograms (AFCL <120 ms; "rapid fires"); and
4. slow nonfractionated electrograms (AFCL >120 ms).

Multipolar electrogram dispersion and non-dispersion regions, illustrate that fractionated electrograms are found in both dispersion and non-dispersion regions.

CFAE software can be used, but CFAE ablation is not guided by the software, but based on visual judgement. Preferably a CFAE map will be made before ablation to judge the sites of most extensive CFAE sites. Baseline mapping in both atria will be performed during AF with the PentaRay multispline catheter sequentially positioned in various regions of the RA and LA. At each location, the catheter will be maintained in a stable position for a minimum of 2.5 s. The operator will look for dispersion areas (electrograms exhibiting both time and spatial dispersion). Where dispersion are found and/or the catheter is not stable for 2.5 s, acquisitions will be repeated.

Additional risks: No additional risks are anticipated for patients enrolled in this study compared to patients undergoing ablation of symptomatic AF outside of the study, because the same catheter is used as in patients outside the study, and both methods (PVI and CFAE) are part of daily practice. Although none reported in the literature so far, CFAE ablation may cause more extensive lesions than other ablation for persistent atrial fibrillation, especially in the posterior wall. This in turn may cause pericardial effusion, myocardial rupture and atrio-esophageal fistula. All of these are potentially life threatening. However, energy settings are changed according to myocardial wall size and pressure recordings, in order to prevent these complications. Furthermore, also in the group of wide antral ablation, the posterior wall is targeted, possibly resulting in the same events. For prevention of posterior wall injury, temperature monitoring in the oesofagus may be used.

Thrombus formation is a complication that can occur with any ablation technique. Thrombi may dislodge and embolize, causing a stroke, myocardial infarction or other ischemic event. Therefore, it is required that activated clotting time (ACT) is kept above 300 seconds. This should be monitored every 30 minutes, and heparin should be administered depending on the outcome. The operator is responsible for maintaining an adequate ACT.

Radiation exposure during the fluoroscopic imaging of the catheters may result in an increase in the lifetime risk of developing a fatal malignancy (0.1%) or a genetic defect in offspring (0.002%).

Potential Benefit: The direct benefit for patients undergoing ablation is the potential elimination of AF episodes. It is furthermore expected that quality of life will improve and less frequent hospitalization will be needed. Whether further morbidity as cerebral vascular events are prevented is subject to discussion. The information gained from the conduct of this study may benefit patients with AF by improving future treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent atrial fibrillation, defined as atrial fibrillation which is:

   1. Sustained beyond 7 days but no more than one year.
   2. Or lasting less than 7 days, but longer than 48 hours and necessitating pharmacologic or electrical cardioversion.
2. Documentation of atrial fibrillation on either a 12-lead ECG or transtelephonic monitoring (TTM), or ambulatory holter monitoring or telemetry strip and a physician's note showing continuous AF.
3. Failure of at least one AAD (Class I or III) as evidenced by recurrent symptomatic AF or intolerable side effects of the AAD.
4. Signed Patient Informed Consent Form.
5. Age 18 years or older.
6. Able and willing to comply with all pre- and follow-up testing and requirements.

Exclusion Criteria:

1. Continuous AF > 12 months (1-Year) (Longstanding Persistent AF).

1. Previous surgical or catheter ablation for atrial fibrillation.
2. Any cardiac surgery within the past 2 months (60 days) (includes PCI).
3. CABG surgery within the past 6 months (180 days).
4. Subjects that have ever undergone valvular cardiac surgical procedure (ie, ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve).
5. Cardioversion refractory (the inability to restore sinus rhythm for 30 secs or longer following electrical cardioversion).

   1. If a patient does not have documented evidence of being successfully cardioverted (NSR > 30 secs), the patient must be cardioverted prior to the ablation procedure with the study catheter.
   2. Failure to cardiovert based on the above criteria is considered a screen failure.
6. Documented LA thrombus on imaging.
7. LA size >50 mm.
8. LVEF < 30%.
9. Contraindication to anticoagulation (heparin or warfarin).
10. History of blood clotting or bleeding abnormalities.
11. Myocardial infarction within the past 2 months (60 days).
12. Documented thromboembolic event (including TIA) within the past 12 months (365 days).
13. Rheumatic Heart Disease.
14. Uncontrolled heart failure or NYHA function class III or IV.
15. Awaiting cardiac transplantation or other cardiac surgery within the next 12 months (365 days).
16. Unstable angina.
17. Acute illness or active systemic infection or sepsis.
18. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
19. Diagnosed atrial myxoma.
20. Presence of implanted ICD.
21. Significant severe pulmonary disease, (eg, restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces chronic symptoms.
22. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
23. Women who are pregnant (as evidenced by pregnancy test if pre- menopausal).
24. Enrollment in an investigational study evaluating another device, biologic, or drug.
25. Presence of intramural thrombus, tumor or other abnormality that precludes vascular access, or manipulation of the catheter.
26. Presence of a condition that precludes vascular access.
27. Life expectancy or other disease processes likely to limit survival to less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-10-12 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Freedom from recorded atrial fibrillation or atrial flutter or atrial tachycardia (>30 seconds) recurrences without the use of class I or III AADs | 18 months
  Freedom from recorded atrial fibrillation or atrial flutter or atrial tachycardia recurrences (>30 seconds) without the use of class I or III AADs through 18 months follow-up, post blanking period after ablation on either a 12 lead ECG on visits or on 24 hour holter monitoring or on symptom-driven event monitoring

SECONDARY OUTCOMES:
Freedom from recorded atrial fibrillation or atrial flutter or atrial tachycardia recurrences (>30 seconds) regardless of antiarrhythmic drugs | 18 months
  Freedom from recorded atrial fibrillation or atrial flutter or atrial tachycardia recurrences (>30 seconds) through 18 months follow-up on either a 12 lead ECG on visits or on 24 hour holter monitoring or on symptom-driven event monitoring, regardless of antiarrhythmic drugs
Freedom from recorded atrial fibrillation or atrial flutter recurrences (>30 seconds) regardless of antiarrhythmic drugs | 18 months
  Freedom from recorded atrial fibrillation or atrial flutter recurrences (>30 seconds) through 18 months follow-up on either a 12 lead ECG on visits or on 24 hour holter monitoring or on symptom-driven event monitoring, regardless of antiarrhythmic drugs
Freedom from recorded atrial fibrillation or atrial flutter or atrial tachycardia recurrences (>30 seconds), without a new AAD or a previously failed AAD at a greater than the highest ineffective historical dose | 18 months
  Freedom from recorded atrial fibrillation or atrial flutter or atrial tachycardia recurrences (>30 seconds) through 18 months follow-up on either a 12 lead ECG on visits or on 24 hour holter monitoring or on symptom-driven event monitoring, without a new AAD or a previously failed AAD at a greater than the highest ineffective historical dose
Freedom from recorded atrial fibrillation (>30 seconds), regardless of antiarrhythmic drugs | 18 months
  Freedom from recorded atrial fibrillation (>30 seconds) through 18 months follow-up on either a 12 lead ECG on visits or on 24 hour holter monitoring or on symptom-driven event monitoring, regardless of antiarrhythmic drugs
Clinical/partial success at 18 months regardless of antiarrhythmic drug use | 18 months
  Clinical/partial success at 18 months regardless of antiarrhythmic drug use, defined as a 75% or greater reduction in the number of AF episodes and/or the duration of AF episodes, or the % time a patient is in AF as assessed with a device capable of measuring AF burden
Time to first symptomatic, recorded AF recurrence | 18 months
  Time to first symptomatic, recorded AF recurrence
Time to first electrocardioversion | 18 months
  Time to first electrocardioversion
Symptoms associated with atrial arrhythmias | 18 months
  Symptoms associated with atrial arrhythmias. Measured by CCS-SAF scale (Canadian Cardiovascular Society Severity of Atrial Fibrillation Scale)
Decreased anti-arrhythmic and/or anticoagulant drug use. | 18 months
  Decreased anti-arrhythmic and/or anticoagulant drug use will be recorded by checking the patients medication chart
Quality of life at 6 and 12 months compared to baseline | 6 months and 12 months
  Quality of life at 6 and 12 months compared to baseline. Measured by SF36-version 2
Number of redo-procedures | 18 months
  Number of redo-procedures
Total time of fluoroscopy | 1 day
  Total time of fluoroscopy
Total procedure time | 1 day
  Total procedure time (minutes from introduction of first catheter to withdrawal of last catheter)
Total ablation time | 1 day
  Total ablation time
Clinical adverse events | 18 months
  Clinical adverse events (TIA,CVA, hemorrhage, tamponade, myocardial infarction, symptomatic pulmonary vein stenosis (> 50%), or other complications associated with AF ablation as listed in and defined by the table 6 of the 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation2)
The combined endpoint consisting of: Mortality and Hospitalization | 18 months
  The combined endpoint consisting of: Mortality and Hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jaap-Jan J. Smit, MD, PhD, Principal Investigator — Isala
Locations (4):
- France (2):
  - Hopital Saint Joseph, Marseille
  - CHU de Nice, Nice
- Kagoshima University, Kagoshima, Japan
- Isala, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seitz J, Bars C, Theodore G, Beurtheret S, Lellouche N, Bremondy M, Ferracci A, Faure J, Penaranda G, Yamazaki M, Avula UM, Curel L, Siame S, Berenfeld O, Pisapia A, Kalifa J. AF Ablation Guided by Spatiotemporal Electrogram Dispersion Without Pulmonary Vein Isolation: A Wholly Patient-Tailored Approach. J Am Coll Cardiol. 2017 Jan 24;69(3):303-321. doi: 10.1016/j.jacc.2016.10.065. PMID 28104073